CLINICAL TRIAL: NCT02491528
Title: A Multi-center, Randomized, Open-label, Parallel-group, Phase Ⅲ Study to Evaluate the Efficacy and Safety of Insulin Aspart Injection in Patients With Diabetes Mellitus Compared to NovoRapid®
Brief Title: A Phase III Study of Insulin Aspart Injection to Evaluate the Efficacy and Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DB021L012015
Record Dates: First submitted 2015-06-05; First posted 2015-07-08 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2015-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin Aspart injection (Experimental): Subcutaneous injection of insulin Aspart prior to three meals every day, while subcutaneous injection of Lantus at bedtime.
  Interventions: Biological: insulin Aspart injection
- insulin Aspart injection (NovoRapid) (Active Comparator): Subcutaneous injection of insulin Aspart (NovoRapid) prior to three meals every day, while subcutaneous injection of Lantus at bedtime.
  Interventions: Biological: insulin Aspart injection (NovoRapid)

INTERVENTIONS:
Biological: insulin Aspart injection — Subcutaneous injection of insulin Aspart prior to three meals every day, while subcutaneous injection of Lantus at bedtime.
  Arms: insulin Aspart injection
Biological: insulin Aspart injection (NovoRapid) — Subcutaneous injection of insulin Aspart injection (NovoRapid) prior to three meals every day, while subcutaneous injection of Lantus at bedtime.
  Arms: insulin Aspart injection (NovoRapid)

SUMMARY:
This is a multicenter, randomized, open, parallel group, active-controlled study. The study period is 25 to 26 weeks, including screening period of 1-2 weeks and treatment period of 24 weeks.

DETAILED DESCRIPTION:
After the screening visit, all patients who met all inclusion criteria and do not meet any of the exclusion criteria were randomized into the experimental group or the controlled group. The subjects in the experimental arm will receive insulin aspart injection combined with basal insulin (Lantus ®), and the subjects in the controlled arm will receive NovoRapid ® (active control) combined with basal insulin (Lantus ®). The experimental drug or the controlled drug will be administered subcutaneously prior to three meals (or can be administered immediately after meal if necessary), and the basal insulin (Lantus ®) will be administered at bedtime. The treatment period is 24 weeks, during which the subjects will be followed up at the clincic cetres at 1, 2, 4, 8, 12, 18, 24 weeks of treatment. At the end of 24-week treatment, if the adverse events continue, the subjects will be followed until recovery or stabilization of the AEs.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed with diabetes；
* BMI≤35.0 kg/m2；
* Insulin therapy for at least 3 months before recruitment；
* HbA1c7~13%

Exclusion Criteria:

* Patients to study drug allergy；
* to Liver and kidney impairment；
* Liver and kidney impairment；
* used systemic steroid treatment in past 2 months .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2016-08-12 (Actual)

PRIMARY OUTCOMES:
The change of relative baseline HbA1c | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: WP Jia, Principal Investigator — The 6th people's hospital of Shanghai
Locations (2):
- China (2):
  - Affiliated hospital of Weifang Medical University, Weifang, Shandong
  - The 6th people's hospital of Shanghai, Shanghai, Shanghai Municipality